CLINICAL TRIAL: NCT05411575
Title: A Randomized, Double-blind, Placebo-controlled, Two Parallel Groups, International Multicenter Trial to Evaluate the Effect of Plerixafor in Acute Respiratory Failure Related to COVID-19.
Brief Title: Plerixafor in Acute Respiratory Distress Syndrome Related to COVID-19 (Phase IIb)
Acronym: LEONARDO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants Enrolled
Sponsor: 4Living Biotech (Industry)
Responsible Party: Sponsor
Organization: 4P-Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4LB-LEO-P
Record Dates: First submitted 2022-05-15; First posted 2022-06-09 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; COVID-19
Keywords: COVID-19; ARDS
MeSH Terms: conditions — COVID-19 | interventions — plerixafor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): continuous intravenous infusion for 7 days of Placebo
  Interventions: Other: Placebo
- Plerixafor (Experimental): Plerixafor (Mozobil®) continuous intravenous infusion for 7 days
  Interventions: Drug: Plerixafor 20 MG/ML [Mozobil]

INTERVENTIONS:
Drug: Plerixafor 20 MG/ML [Mozobil] — Plerixafor (Mozobil®) continuous intravenous infusion for 7 days
  Arms: Plerixafor
Other: Placebo — Placebo continuous intravenous infusion for 7 days
  Arms: Placebo

SUMMARY:
This phase IIb study, LEONARDO is a multicenter, randomized, double-blind, placebo- controlled, parallel group study, to assess the therapeutic efficacy and safety of Plerixafor in patients over 18 years of age,

* with acute respiratory failure related to COVID-19 and
* Recently admitted in ICU or equivalent structure (within 48 hours) for COVID-19 related respiratory failure
* without invasive mechanical ventilation and
* requiring oxygen support ≥ 5L/min to obtain a transcutaneous O2 saturation > 94% A total of 150 participants, will be randomized in a 2:1 ratio to receive either Plerixafor (n=100) or placebo (n=50) as a continuous IV infusion for 7 days (from D1 to D8) in addition to standard of care (e.g. glucocorticoids...).

Safety data will be reviewed by an independent Data and Safety Monitoring Board (DSMB) during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age,
* Using contraceptive consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Willing and able to provide written informed consent (or provided by legally acceptable representative if he/she is present and if in line with local regulations),
* Admitted in ICU within 48 hours before randomization for COVID-19 related respiratory failure. (ICU or equivalent medical structure according to country specificities e.g., Acute Respiratory Care Unit, High Dependency Care Unit if they can provide: continuous IV infusion,continuous ECG, respiratory rate, percutaneous oxygen saturation screen monitoring, high flow nasal oxygen)
* Not requiring immediate (within 24-36 hours) invasive mechanical ventilation according to investigator's judgment,
* Confirmed pneumoniae due to SARS-CoV-2, Laboratory-confirmed SARS-CoV-2 infection as determined by RT-PCR (in nasopharynx or throat samples) or other commercial or public health assay in any specimen, performed within 2 weeks prior to randomization,
* Acute respiratory failure requiring oxygen support (≥ 5L/min) to achieve a transcutaneous oxygen saturation > 94%,
* Estimated glomerular filtration rate (eGFR) > 50 mL/min/1.73m2 by the CKD-EPI (Chronic Kidney Disease - Epidemiology Collaboration) equation.

Exclusion Criteria:

* Pregnancy or breast feeding,
* Anticipated transfer to another hospital, which is not a study site within 72 hours of randomisation,
* Need for Invasive mechanical ventilation at time of inclusion,
* Evidence of uncontrolled bacterial pneumopathy or active infection other than SARS-Cov-2 (laboratory confirmation),
* Primitive pulmonary arterial hypertension,
* Cardio-vascular co-morbidity:

  * History of vascular ischemic events (myocardial infarction or stroke) or congestive heart failure or peripheral arterial disease,
  * History or current significant cardiac rhythm disorders (e.g., ventricular tachycardia),
  * Known medical history of proven symptomatic postural hypotension,
* Known cancer (solid or blood) in the last 5 previous years or previous haematological disorders (malignancies and other chronic conditions) or having received bone marrow transplant,
* Inadequate haematological function defined by:

  * Neutrophil count < 1.0 x 109/L,
  * Haemoglobin < 9.0 g/dL (90 g/L),
  * Platelets < 100 x 109/L,
* Kaliemia < 3.5 mmol/L and/or total Calcemia < 2.2 mmol/L,
* Inadequate hepatic function defined by Aspartate aminotransferase (AST) and/or Alanine Aminotransferase (ALT) > 3 x upper limit of normal (ULN) and/or Total bilirubin > 2 x ULN,
* Patients with known allergy to Plerixafor or its excipients.
* Previous (within 4 weeks) or current participation in another clinical study other than an observational study.
* Patients with auto immune disease treated or not,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-19 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that Plerixafor is able to reduce the need for invasive mechanical ventilation or death in severe COVID-19 patients admitted in Intensive Care Unit (ICU) | Day 1- Day 28
  Proportion of patients with need for invasive mechanical ventilation or death between randomization and D28

SECONDARY OUTCOMES:
To evaluate the efficacy of Plerixafor compared to placebo on Mortality between randomization and D28 | Day 1-Day 28
  Percentage of death (all-cause mortality)
To evaluate the efficacy of Plerixafor compared to placebo on Mortality between randomization and D90 | Day 1-Day 90
  Percentage of death (all-cause mortality)
To evaluate the efficacy of Plerixafor compared to placebo on Ventilator-free days between randomization and D28 | Day 1-Day 28
  Number of Ventilator-free days
To evaluate the efficacy of Plerixafor compared to placebo on Duration of mechanical ventilation between randomization and D90 | Day 1-Day 90
  Duration of invasive mechanical ventilation in survivors
To evaluate the efficacy of Plerixafor compared to placebo on Length of ICU stay between randomization and D90 | Day 1-Day 90
  Number of ICU stay days
To evaluate the efficacy of Plerixafor compared to placebo on Respiratory function including FEV1, FVC, PaO2 and Transfer Lung Capacity for carbon monoxide (TLCO), 6-minute walk test | Day 1-Day 90
  Respiratory function at 3 months (FEV-1, FVC, PaO2, TLCO, 6-minute walk test)
To evaluate the efficacy of Plerixafor compared to placebo on Clinical improvement | Day 1, Day 8, Day 14 Day 28, Day 90
  Ordinal Scale for Clinical Improvement (Clinical improvement: 7-point ordinal scale of the WHO Master Protocol (WHO, 2020). 1: not hospitalized up to 7:death)
To evaluate the efficacy of Plerixafor compared to placebo on Level of consciousness | Day 1-Day 8, Day 14, Day 28, Day 90
  Level of consciousness (Alert, Voice, Pain, Unresponsive scale)
To evaluate the efficacy of Plerixafor compared to placebo on SpO2 status | Day 1-Day 8, Day 14, Day 28, Day 90
  Measure of SpO2 via pulse oxymetry
To evaluate the efficacy of Plerixafor compared to placebo on Respiratory/oxygenation status | Day 1-Day 8, Day 14, Day 28, Day 90
  Measure of Partial pressure of oxygen (PaO2), Partial pressure of carbon dioxide (PaCO2), Bicarbonate (HCO3),
To evaluate the efficacy of Plerixafor compared to placebo on CRP, fibrinogen and D-dimers levels | Day 1, Day 3, Day 8, Day 14, Day 28
  Blood CRP, fibrinogen, D-dimers levels
To evaluate the efficacy of Plerixafor compared to placebo on Safety AEs | up to Day 90
  Incidence of treatment-emergent AEs (TEAEs), serious AEs (SAEs), and AEs of special interest (AESIs), incidence of treatment on discontinuation and withdrawals due to TEAEs
To evaluate the efficacy of Plerixafor compared to placebo on Safety/Lab tests | up to Day 90
  Quantification of White Blood Cells count and differential, Red Blood Cells count, hemoglobin level, Mean Corpuscular Volume, Reticulocyte and Platelet counts . Blood Chemistry (Creatinine, AST, ALT, total bilirubin, Potassium, total Calcium)

CONTACTS AND LOCATIONS:
Locations (14):
- Bulgaria (9):
  - Multiprofile Hospital for Active Treatment AD Haskovo, Haskovo
  - Multiprofile Hospital For Active Treatment Pazardzhik AD, Pazardzhik
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - Multiprofile Hospital for Active Treatment Dr Ivan SeliminskiSliven AD, Sliven
  - University First Multiprofile Hospital for Active Treatment Sofia St John the Baptist, Sofia
  - Military Medical Academy Multiprofile Hospital for Active Treatment Sofia, Sofia
  - University Hospital for Active Treatment and Emergency Medicine NI Pirogov EAD, Sofia
  - MHAT Sveta Anna Sofia AD, Sofia
  - University Multiprofile Hospital for Active Treatment Prof Dr Stoyan Kirkovich AD, Stara Zagora
- France (5):
  - Centre Hospitalier d'Argenteuil, Argenteuil
  - Hôpital Saint André, Bordeaux
  - Centre Hospitalier Départemental de Vendée - Les Oudairies, La Roche-sur-Yon
  - Hôpital Haut-Lévêque, Pessac
  - Hôpital Civil de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided